CLINICAL TRIAL: NCT06659471
Title: A Three-Month Bleeding Model Clinical Study
Brief Title: Brief Title: a Clinical Study to Assess Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021117
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2022-03

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 0.76% Sodium Monofluorophosphate (Sham Comparator): 0.76% Sodium Monofluorophosphate
  Interventions: Drug: 0.76% Sodium Monofluorophosphate Dentifrice
- 0.454% Stannous Fluoride (Active Comparator): 0.454% Stannous Fluoride
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice
- 0.454% Stannous Fluoride, 4.7 pH (Experimental): 0.454% Stannous Fluoride, 4.7 pH
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice
- 0.454% Stannous Fluoride, 5.8 pH (Experimental): 0.454% Stannous Fluoride, 5.8 pH
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice

INTERVENTIONS:
Drug: 0.76% Sodium Monofluorophosphate Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: 0.76% Sodium Monofluorophosphate
Drug: 0.454% Stannous Fluoride Dentifrice — Whole mouth brushing with a toothpaste, twice daily for the duration of the study.
  Arms: 0.454% Stannous Fluoride; 0.454% Stannous Fluoride, 4.7 pH; 0.454% Stannous Fluoride, 5.8 pH

SUMMARY:
The objective of this learning clinical study is to evaluate the effects of formulation chemistry on gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be in general good health as determined by the Investigator based on a review of the health history/update for participation in the trial;
* Have at least 20 gradable teeth;
* Have established gingivitis with 10-70 % bleeding sites;
* Agree to return for scheduled visits and follow the study procedures;
* Agree to refrain from use of any non-study oral hygiene products for the duration of the study;
* Agree to delay any elective dentistry, including dental prophylaxis, until the completion of the study.

Exclusion Criteria:

* Having taken medications (antibiotic, anti-inflammatory, or anti-coagulant) which could alter gingival bleeding within 4 weeks of the Baseline Visit;
* Having any oral conditions that could interfere with study compliance and/or examination procedures, such as widespread caries, soft or hard tissue tumor of the oral cavity, or advanced periodontal disease;
* Having known hypersensitivity to the test products;
* Having removable oral appliances;
* Having fixed facial or lingual orthodontic appliances;
* Self-reported pregnancy or lactation;
* Having any diseases or condition that might interfere with the safe participation in the study;
* Having an inability to undergo study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Number Bleeding Sites | 3 months, 1 month
  Number of bleeding sites derived from the Löe-Silness Gingivitis Evaluation based on a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).

SECONDARY OUTCOMES:
Löe-Silness Gingivitis Evaluation | 3 months, 1 month
  Löe-Silness Gingivitis Evaluation is a validated assessment of gingival health looking at inflammation and bleeding based on a 4 point range 0 (normal gingiva) to 3 (severe inflammation).

CONTACTS AND LOCATIONS:
Locations (1):
- Silverstone Research, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No